CLINICAL TRIAL: NCT01307410
Title: A Comprehensive Longitudinal Cohort Study in Type 2 Diabetes With High Risk of Cardiovascular Diseases in China - 3B Extension A Study of China Cardiometabolic Registries (CCMR)
Brief Title: A Comprehensive Longitudinal Cohort Study in Type 2 Diabetes With High Risk of Cardiovascular Diseases in China
Acronym: CCMR-3B Ext
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Cardiometabolic Registries (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry); VitalStrategic Research Institute (Other); China Gerontological Society (Other); Chinese Medical Doctor Association (Other)
Responsible Party: Sponsor
Other Study IDs: CCMR-303-3B Extension
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes
Keywords: Patients with type 2 diabetes and participated in 3B Study
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with CAD: Patients with hypertension and dyslipidemia with prior CAD
- without CAD: Patients with hypertension and dyslipidemia without prior CAD

SUMMARY:
In 2010, the sponsor conducted an observational study, entitled as "Nationwide Assessment of Cardiovascular Risk Factors: Blood Pressure, Blood Lipid, and Blood Glucose, in Chinese Patients with Type 2 Diabetes - 3B Study " which was to evaluate the level of cardiovascular diseases (CVD) risk factor control and its regional difference in China. As a continuation, this extension of the 3B Study is designed to assess the incidence of cardiovascular events, cardio-renal events, and other microvascular complications, in 1, 2 and 3 years in patients with type 2 diabetes and with high risk of (CVD) with or without existing or history of coronary artery diseases.

DETAILED DESCRIPTION:
Limited by its cross sectional design, 3B study was not be able to provide any information on how various patterns of treatment and prescribing behaviors would impact the outcomes of prevention of cardiovascular and cardio-renal diseases in type 2 diabetes longitudinally. This information, however, would be crucial in better guiding the real world medical practice and maximizing the effectiveness of medical treatment for better controlling cardiovascular risk factors.

The 3B Extension study is thus designed to extend the 3B study by continuing to follow up on enrolled patients for 3 years. The 3B Extension study is expected to demonstrate the clinical outcomes of nationally representative type 2 diabetes patients who are treated by endocrinologists, cardiologists and nephrologists separately in all tiers of hospitals, as measured by diabetes progression, incidence of cardiovascular complications, and incidence of microvascular complications. It will be the first study of this scale in China based on its exclusivity, extensiveness, and the level of government and national thought leaders' support. It will be conducted in collaboration with the advisory board of China Cardiometabolic Registries (CCMR).

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Outpatients who meet the inclusion and exclusion criteria of 3B study
* With hypertension,dyslipidemia and one of the following:
* History of acute coronary artery disease or ischemic stroke
* Age > 65 years old
* Overweight or obesity (BMI > 24 kg/m2)
* Microalbuminuria or albuminuria
* Current smoker

Exclusion Criteria:

* Patients with type 1 DM
* Pregnant or breast feeding women
* Patients who are unable to or not willing to return for follow up visits every 6 months for 3 years;
* Patients have severe heart failure (NYHA Class III-IV)
* Patients with severe renal deficiency (creatinine clearance < 30 ml/min)
* Patients who are not willing to sing the informed consent form;
* Patients who are participating in any other interventional clinical studies,

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes who previously participated in the 3B study from either community (tier 1), regional (tier 2), or teriary (tier 3) hospitals
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of CVD events | 3 years
  The CVD event is defined as composite of :
  * Acute myocardial infarction
  * Stroke
  * Cardiovascular death

SECONDARY OUTCOMES:
Annual incidence of microvascular complications | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, MD, Principal Investigator — People's Hospital, Beijing University; Dayi Hu, MD, Principal Investigator — People's Hospital, Beijing University

REFERENCES:
- See also: Website for China Cardiometabolic Registries — http://www.CCMRegistry.org